CLINICAL TRIAL: NCT03721588
Title: Evaluation of Clinical and Suicidal Behavior Characteristics Among Urban, Turkish Middle-Age Depressive Patients With Comorbid Adult Attention Deficit Hyperactivity Disorder
Brief Title: Clinical and Suicidal Features of Urban, Turkish Middle Age Depressive Patients With Comorbid ADHD
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esin Erdoğan, Psychiatry Department, MD, Bozyaka Training and Research Hospital
Other Study IDs: dresinerdogan
Record Dates: First submitted 2018-10-12; First posted 2018-10-26 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Depressive Disorder, Major; Adult Attention Deficit Hyperactivity Disorder; Suicide
MeSH Terms: conditions — Depressive Disorder, Major; Attention Deficit Disorder with Hyperactivity; Suicide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major depressive disorder: MDD; patients with diagnosis of major depressive disorder, Clinical interviews, psychometric scales were applied.
  Interventions: Other: Clinical interviews, psychometric scales were applied.
- MDD and ADHD: MDD; major depressive disorder ADHD; attention deficit hyperactivity disorder, Clinical interviews, psychometric scales were applied.
  Interventions: Other: Clinical interviews, psychometric scales were applied.

INTERVENTIONS:
Other: Clinical interviews, psychometric scales were applied.

SUMMARY:
In the presence of attention deficit hyperactivity disorder (ADHD) together with additional psychiatric diseases, the treatment process and prognosis of both ADHD and psychiatric comorbidity are adversely affected. The aim of this study is to compare the characteristics concerning the suicidal behavior of the patients with major depressive disorder (MDD) who have (ADHD+) or do not have (ADHD-) adult ADHD comorbidity and their responses to depression treatment. 96 inpatients were included in the study. Socio-demographic data form, Hamilton Depression Scale (HDRS), Wender Utah Rating Scale (WURS), Adult ADD/ADHD DSM IV- Based Diagnostic Screening and Rating Scale (A-ADHD), Personal and Social Performance Scale (PSP) were applied to the cases. In the study, depression starts at an early age in individuals with comorbid ADHD and the depression treatment progress changes negatively. This group of patients is at greater risk in terms of suicidal behavior. For these reasons, clinicians should be careful during ADHD and depression management in adults.

DETAILED DESCRIPTION:
Suicidal behavior is a serious cause of mortality and morbidity in terms of psychiatric diseases. Suicidal ideation and suicide attempts that do not result in death cause many social and emotional problems, but they are the most important risk factors for the next suicide attempt and death resulting from suicide.[1,2] It has been reported that 90% of the completed suicide attempt cases are accompanied by a psychiatric disease and depressive disorders are seen at a highest level. [3] Attention-deficit hyperactivity disorder (ADHD) is a neurodevelopmental disorder with symptoms of inattention, hyperactivity and impulsivity that is seen as of childhood.[4-6] ADHD disrupts the individuals' functionality in many fields such as academic, social and business life.[7] It also increases the risk of comorbidity of many psychiatric diseases.[8-10] In the studies carried out, it has been reported that depression is seen in rates ranging from 16% to 31% in cases with adult ADHD [11] and it was accompanied by ADHD in 15% of cases with depression.[12] In depressive adults with ADHD comorbidity, resistance to depression treatment develops and the longitudinal progress of both diseases is adversely affected.[13-14] In the literature review, it has been reported that suicide risk increased in children,[15] in university students,[16] in young women,[17] in ADHD and depression comorbidity and the clinical progress of depression was adversely affected.[18] Studies examining the relationship of suicide in ADHD and depression comorbidity in adults have been mostly carried out in young adults and it has been suggested by researchers to investigate the association of ADHD and depression in older adults.[19-22] The aim of this study was to compare the suicidal behavior, the onset age of depression and the respond to the treatment of the depressive disorder inpatients in the psychiatry service who are with and without comorbid ADHD. Hypothesis of this study is that the following will be observed in the adult depression patients with ADHD comorbidity; depression starting at an earlier age, having much more suicide attempts (number of suicide attempts in the past) that are much serious (requiring medical treatment) and having more severe depression (depression scale scores) and worse self-functionality during discharge from the hospital.

Material & Methods Complying with DSM-IV criteria and Hamilton Depression Scale (HDRS) being over 16 points during hospitalization have been determined to be the criteria for inclusion in the research. In total, 96 patients were included in the study. All cases were interviewed with the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I).[23] Other comorbid psychiatric disorders were excluded. Adult ADHD diagnosis has been confirmed by two different researchers for each case (DHD, EE). In the retrospective investigation of ADHD diagnosis, cases who got the score of 36 and above in the Wender Utah Rating Scale (WURS) have been included in the study.

Investigators evaluated suicidal behavior in a similar manner to the methods used in some previous studies.[20,24,25] In the sociodemographic data form, suicidal ideation in the past (Have you ever thought about ending your life before? / Yes or No), suicide attempt (Have you ever attempted suicide before? / Yes or No) and number of suicide attempts have been recorded. Material

Socio-demographic data form:

Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) [26] Hamilton Depression Rating Scale (HDRS): [28] Adult ADD/ADHD DSM IV- Based Diagnostic Screening and Rating Scale (A-ADHDS) has been developed by Atilla Turgay in Canada.[29,30] Wender Utah Rating Scale (WURS): [31,32] Personal and Social Performance Scale (PSP): [33,34] Statistical analysis: SPSS Statistics Version 22.0 has been used for data analysis. The distribution characteristics of the variables have been evaluated by using the Shapiro-Wilk test. Student-t test has been used to compare normal distribution parameters and Mann-Whitney U test has been used for abnormal distribution parameters. According to the ADHD comorbidity, suicide attempt has been compared with the Pearson chi-squared test. P values below 0.05 have been considered to be statistically significant results.

Results The mean age of the patients was 39.1±10.4. 57% (n=55) of all patients were females. 31% (n=30) were single / never married, 53% (n=49) were married / living with a spouse, 16% (n=17) were divorced or living apart There was no statistically significant difference found between patients with ADHD comorbidity (ADHD+) and patients with only MDD (ADHD-) in terms of gender, age, marital status and education.

In the ADHD+ group, depression started at an earlier age than the ADHD- group (p= .011). The average HDRS scores during admission to hospital and discharge from the hospital were significantly higher in the ADHD+ group (p<.000). Moreover, the average PSP scores of the ADHD+ group at admission to hospital was lower than the ADHD- group and there was a statistically significant difference between them (p = .002). There was no difference between the groups during their discharge with regards to PSP scores (p = .46).

Suicidal ideation (p = .018) and suicide attempts (p = .013) throughout life were higher in the ADHD+ group than the ADHD- group. In the ADHD+ group, the rate of suicide attempts that require medical intervention was higher (p = .001). A comparison of the suicidal behavior characteristics of ADHD+ and ADHD- groups is presented in Table 3 and it has been shown graphically whether the cases have attempted suicide according to ADHD comorbidity throughout their lives.

Discussion n ADHD+ group, depression has started at an earlier age, the severity of depression has been higher during discharge from the hospital and suicidal ideation, number of suicide attempts and suicide attempts requiring medical intervention throughout their lives were found to be high. Depressive disorder patients with ADHD comorbidity in our study have got their first depression diagnosis at an early age. Similar results have been found by other researchers.[17,35, 36] Another result of study was that the discharge HDRS scores of the depressive patients with ADHD comorbidity were higher. Resistance to depression treatment has been reported in the association of ADHD and depression.[38,39] ADHD causes disruptions of the individuals' functionality in many areas of their lives starting from childhood [40,41] and it has also been reported that there is a decrease in social skills and self-esteem of adolescents with ADHD.[42] It has been suggested that in the event of frequent recurrent depressive attacks, inability of remission, continuation of residual symptoms and inadequate response to classical therapies of cases with depression, a retrospective investigation of ADHD[38,39] and treatment planning for ADHD should be made.[18,36,43] As a result of the study, the rate of suicidal ideation throughout life and number of suicide attempts were found to be higher in ADHD+ group. As mentioned literature, 90% of the cases who attempted suicide are accompanied by a psychiatric disorder where depressive disorder is the most common one.[3] It has been reported that suicide attempts are related to depression duration or impulsivity.[43] In addition, as a result of the research, in the association of ADHD and depression, the number of suicidal behaviors that are serious enough to require medical care is also higher. This finding has also been reported by other researchers when literature is evaluated.[16,25] In adults, suicide is more common in ADHD and MDD comorbidity and suicidal attempts may lead to more dangerous consequences (such as being in the intensive care unit, causing disability).

ELIGIBILITY:
Inclusion Criteria:

1. Complying with DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth) criteria for major depression
2. Hamilton Depression Scale (HDRS) being over 16 points during hospitalization

Exclusion Criteria:

1. Mental retardation
2. Psychotic disorder
3. Alcohol or substance addiction
4. History of head trauma
5. Being under psychostimulant treatment

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: inpatiets with diagnosis of major depressive disorder
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
depressive inpatients with comorbid ADHD (n=48) and without comorbid ADHD (n=48) were compared according to the suicidal behavior, the onset age of depression, the response to the treatment, and psychosocial functioning. | 2 years
  Clinical interviews, psychometric scales such as, Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I), Hamilton Depression Rating Scale (HDRS), Adult ADD/ADHD DSM IV- Based Diagnostic Screening and Rating Scale (A-ADHDS), Wender Utah Rating Scale (WURS), Personal and Social Performance Scale (PSP) were applied. 96 inpatients were included in the study. In our study, depression starts at an early age in individuals with comorbid ADHD and the depression treatment progress changes negatively. This group of patients is at greater risk in terms of suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Erdogan, MD, Principal Investigator — Bozyaka Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duran S, Fistikci N, Keyvan A, Bilici M, Caliskan M. [ADHD in adult psychiatric outpatients: prevalence and comorbidity]. Turk Psikiyatri Derg. 2014 Summer;25(2):84-93. Turkish. PMID 24936755
- [Result] Agosti V, Chen Y, Levin FR. Does Attention Deficit Hyperactivity Disorder increase the risk of suicide attempts? J Affect Disord. 2011 Oct;133(3):595-9. doi: 10.1016/j.jad.2011.05.008. Epub 2011 Jun 11. PMID 21658780
- [Result] Tamam L, Demirkol ME. Adult attention deficit/hyperactivity disorder and mood disorders. Turkiye Klin J Psychiatry-Special Top 2012;5:48-3.
- [Result] Ekinci S, Öncü B, Canat S. Adult attention deficit hyperactivity disorder: comorbidity and functioning. Anadolu Psikiyatr Derg 2011;12:185-1.